CLINICAL TRIAL: NCT02985801
Title: Pancreatic Enzyme Replacement Therapy (PERT) for Treatment of Exocrine Pancreatic Insufficiency in Patients With Unresectable Pancreatic Cancer
Brief Title: PERT for Treatment of Exocrine Pancreatic Insufficiency in Patients With Unresectable Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to difficulty in recruiting subjects.
Sponsor: Massimo Raimondo, M.D. (Other)
Collaborators: Digestive Care, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Massimo Raimondo, M.D., Professor, College of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-008713
Record Dates: First submitted 2016-11-28; First posted 2016-12-07 (Estimated); Results first posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: Pancreatic Insufficiency; Pancreatic Cancer; Pancreatic Enzyme Abnormality
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Pancreatic Neoplasms | interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo First, then Pancrelipase (Experimental): Placebo oral capsule: 3 capsules taken with or after meals, and 2 capsules taken with or after snacks during 4 weeks in first intervention period, and Pancrelipase 3 capsules are taken with or after meals (4800 lipase units) and 2 capsules with or after snacks (3200 lipase units) during 4 weeks in second intervention period (after 2 week washout period).
  Interventions: Drug: Pancrelipase; Drug: Placebo Oral Capsule
- Pancrelipase First, then Placebo (Experimental): Pancrelipase 3 capsules are taken with or after meals (4800 lipase units) and 2 capsules with or after snacks (3200 lipase units) during 4 weeks in first intervention period, and Placebo oral capsule: 3 capsules taken with or after meals, and 2 capsules taken with or after snacks during 4 weeks in second intervention period (after 2 week washout period).
  Interventions: Drug: Pancrelipase; Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Pancrelipase — Lipase 16,000 United States Pharmacopoeia (USP) units, protease 57,500 USP units, and amylase 60,500 USP units
  Other Names: Pertzye
Drug: Placebo Oral Capsule — Placebo Oral Capsule

SUMMARY:
Does pancreas enzyme replacement (PERT) decrease weight loss and improve quality of life in patients with unresectable pancreatic cancer?

DETAILED DESCRIPTION:
Randomized, double-blind clinical trial aiming to assess the impact of pancreas enzyme replacement therapy in weight loss and quality of life.

Prevalence of pancreatic exocrine insufficiency (PEI) will be determined with fecal elastase-1 test (FE1) in patients with unresectable pancreatic cancer, without evidence of pancreatic duct (PD) or common bile duct (CBD) obstruction based on MRI or / and endoscopic ultrasound (EUS).

Patients with PEI (FE1 <200) receive Pertzye or placebo in a cross-over fashion, each for 4 weeks.

Body weight, body mass index (BMI), body composition (Bioimpedance), are measured at the time of diagnosis of PEI and at 4 and 10 weeks of cross-over treatment. Baseline measurement of Vitamin D-25, Vitamin A, iron (ferritin, total iron binding capacity (TIBC), iron), Vitamin B12,Tissue transglutaminase IgA (tTG) with total Immunoglobulin A (IgA).

Quality of Life (pain, diarrhea, weight, bloating, etc.) assessed at 0,4,10 weeks with the Functional Assessment of Cancer Therapy for patients with liver, bile duct and pancreas cancer (FACT-Hep) for physical, social, emotional, and functional quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-80 years
* Underlying pancreatic adenocarcinoma, unresectable (local invasion or distant metastasis)
* On established chemotherapy regimen for pancreas cancer, which will be continued over the time of study
* Fecal elastase-1 test (FE1) less than 200 mcg pancreatic elastase/g stool

Exclusion Criteria:

* Common bile duct obstruction resulting in obstructive jaundice
* Celiac disease
* Crohn's disease
* Benign pancreatic conditions
* Bowel obstruction
* Surgically altered bowel anatomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Raimondo, MD, Principal Investigator — Professor of Medicine
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heffernan N, Cella D, Webster K, Odom L, Martone M, Passik S, Bookbinder M, Fong Y, Jarnagin W, Blumgart L. Measuring health-related quality of life in patients with hepatobiliary cancers: the functional assessment of cancer therapy-hepatobiliary questionnaire. J Clin Oncol. 2002 May 1;20(9):2229-39. doi: 10.1200/JCO.2002.07.093. PMID 11980994
- [Background] Perez MM, Newcomer AD, Moertel CG, Go VL, Dimagno EP. Assessment of weight loss, food intake, fat metabolism, malabsorption, and treatment of pancreatic insufficiency in pancreatic cancer. Cancer. 1983 Jul 15;52(2):346-52. doi: 10.1002/1097-0142(19830715)52:23.0.co;2-z. PMID 6305473
- [Background] Partelli S, Frulloni L, Minniti C, Bassi C, Barugola G, D'Onofrio M, Crippa S, Falconi M. Faecal elastase-1 is an independent predictor of survival in advanced pancreatic cancer. Dig Liver Dis. 2012 Nov;44(11):945-51. doi: 10.1016/j.dld.2012.05.017. Epub 2012 Jun 28. PMID 22749648
- [Background] Sikkens EC, Cahen DL, de Wit J, Looman CW, van Eijck C, Bruno MJ. A prospective assessment of the natural course of the exocrine pancreatic function in patients with a pancreatic head tumor. J Clin Gastroenterol. 2014 May-Jun;48(5):e43-6. doi: 10.1097/MCG.0b013e31829f56e7. PMID 24717227
- [Background] Dutta SK, Rubin J, Harvey J. Comparative evaluation of the therapeutic efficacy of a pH-sensitive enteric coated pancreatic enzyme preparation with conventional pancreatic enzyme therapy in the treatment of exocrine pancreatic insufficiency. Gastroenterology. 1983 Mar;84(3):476-82. PMID 6549746
- [Background] Valerio D, Whyte EH, Schlamm HT, Ruggiero JA, Blackburn GL. Clinical effectiveness of a pancreatic enzyme supplement. JPEN J Parenter Enteral Nutr. 1981 Mar-Apr;5(2):110-4. doi: 10.1177/0148607181005002110. PMID 7195437
- [Background] Bruno MJ, Haverkort EB, Tijssen GP, Tytgat GN, van Leeuwen DJ. Placebo controlled trial of enteric coated pancreatin microsphere treatment in patients with unresectable cancer of the pancreatic head region. Gut. 1998 Jan;42(1):92-6. doi: 10.1136/gut.42.1.92. PMID 9505892
- [Background] Delchier JC, Vidon N, Saint-Marc Girardin MF, Soule JC, Moulin C, Huchet B, Zylberberg P. Fate of orally ingested enzymes in pancreatic insufficiency: comparison of two pancreatic enzyme preparations. Aliment Pharmacol Ther. 1991 Aug;5(4):365-78. doi: 10.1111/j.1365-2036.1991.tb00040.x. PMID 1777547
- [Background] Ghaneh P, Neoptolemos JP. Exocrine pancreatic function following pancreatectomy. Ann N Y Acad Sci. 1999 Jun 30;880:308-18. doi: 10.1111/j.1749-6632.1999.tb09534.x. PMID 10415875
- [Background] DiMagno EP, Malagelada JR, Go VL. The relationships between pancreatic ductal obstruction and pancreatic secretion in man. Mayo Clin Proc. 1979 Mar;54(3):157-62. PMID 431121
- [Background] Graham DY. An enteric-coated pancreatic enzyme preparation that works. Dig Dis Sci. 1979 Dec;24(12):906-9. doi: 10.1007/BF01311943. PMID 510089
- [Background] Halgreen H, Pedersen NT, Worning H. Symptomatic effect of pancreatic enzyme therapy in patients with chronic pancreatitis. Scand J Gastroenterol. 1986 Jan;21(1):104-8. doi: 10.3109/00365528609034631. PMID 3633631
- [Background] Lankisch PG, Lembcke B, Goke B, Creutzfeldt W. Therapy of pancreatogenic steatorrhoea: does acid protection of pancreatic enzymes offer any advantage? Z Gastroenterol. 1986 Dec;24(12):753-7. PMID 3548109
- [Background] Schneider MU, Knoll-Ruzicka ML, Domschke S, Heptner G, Domschke W. Pancreatic enzyme replacement therapy: comparative effects of conventional and enteric-coated microspheric pancreatin and acid-stable fungal enzyme preparations on steatorrhoea in chronic pancreatitis. Hepatogastroenterology. 1985 Apr;32(2):97-102. PMID 2408983
- [Background] Nouisa-Arvanitakis S, Stapleton FB, Linshaw MA, Kennedy J. Therapeutic approach to pancreatic extract-induced hyperuricosuria in cystic fibrosis. J Pediatr. 1977 Feb;90(2):302-5. doi: 10.1016/s0022-3476(77)80657-4. PMID 830926
- [Background] Gullo L, Pezzilli R, Gaiani S. Tolerability and safety of the long-term administration of pancreatic extracts. Pancreas. 1997 Mar;14(2):210-2. doi: 10.1097/00006676-199703000-00018. No abstract available. PMID 9057197
- [Background] Seiler CM, Izbicki J, Varga-Szabo L, Czako L, Fiok J, Sperti C, Lerch MM, Pezzilli R, Vasileva G, Pap A, Varga M, Friess H. Randomised clinical trial: a 1-week, double-blind, placebo-controlled study of pancreatin 25 000 Ph. Eur. minimicrospheres (Creon 25000 MMS) for pancreatic exocrine insufficiency after pancreatic surgery, with a 1-year open-label extension. Aliment Pharmacol Ther. 2013 Apr;37(7):691-702. doi: 10.1111/apt.12236. Epub 2013 Feb 5. PMID 23383603
- [Background] Ramesh H, Reddy N, Bhatia S, Rajkumar JS, Bapaye A, Kini D, Kalla M, Thorat V. A 51-week, open-label clinical trial in India to assess the efficacy and safety of pancreatin 40000 enteric-coated minimicrospheres in patients with pancreatic exocrine insufficiency due to chronic pancreatitis. Pancreatology. 2013 Mar-Apr;13(2):133-9. doi: 10.1016/j.pan.2013.01.009. Epub 2013 Feb 5. PMID 23561971
- [Background] Gubergrits N, Malecka-Panas E, Lehman GA, Vasileva G, Shen Y, Sander-Struckmeier S, Caras S, Whitcomb DC. A 6-month, open-label clinical trial of pancrelipase delayed-release capsules (Creon) in patients with exocrine pancreatic insufficiency due to chronic pancreatitis or pancreatic surgery. Aliment Pharmacol Ther. 2011 May;33(10):1152-61. doi: 10.1111/j.1365-2036.2011.04631.x. Epub 2011 Mar 21. PMID 21418260
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo First, Then Pancrelipase | Pancrelipase First, Then Placebo
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First, Then Pancrelipase | Pancrelipase First, Then Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (7.6) | 68.3 (6.9) | 65.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Body weight will be measured at the time of accrual, and at 4 and 10 weeks of cross-over treatment.
Time Frame: Baseline, 4 weeks, 10 weeks
Population: Study was terminated due to difficulty in recruiting subjects. Data was not collected or analyzed.
Groups:
- Placebo: Subjects who received placebo oral capsule in either the first or last 4 weeks of the study
- Pancrelipase: Subjects who received Pancrelipases oral capsules in either the first or last 4 weeks of the study
Arm/Group | Placebo | Pancrelipase
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Quality of Life Score as Measured by FACT-Hep Scale at 4 Weeks
Description: Quality of life will be measured using the FACT-Hep questionnaire (Functional Assessment of Cancer Therapy for patients with liver, bile duct and pancreas cancer) for physical, social, emotional, and functional quality of life at the time of accrual, and at 4 weeks of cross-over treatment. The FACT-Hep scale consists of 45 questions, with possible responses ranging from 0 (not at all) to 4 (very much). Therefore, the total score can range from 0 (not at all - no issues) to 180 (very much - very poor quality of life).
Time Frame: Baseline, 4 weeks
Population: Study was terminated due to difficulty in recruiting subjects. Data was not collected or analyzed.
Arm/Group | Placebo | Pancrelipase
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Quality of Life Score as Measured by FACT-Hep Scale at 10 Weeks
Description: Quality of life will be measured using the FACT-Hep questionnaire (Functional Assessment of Cancer Therapy for patients with liver, bile duct and pancreas cancer) for physical, social, emotional, and functional quality of life at the time of accrual, and at 10 weeks of cross-over treatment. The FACT-Hep scale consists of 45 questions, with possible responses ranging from 0 (not at all) to 4 (very much). Therefore, the total score can range from 0 (not at all - no issues) to 180 (very much - very poor quality of life).
Time Frame: Baseline, 10 weeks
Population: Study was terminated due to difficulty in recruiting subjects. Data was not collected or analyzed.
Arm/Group | Placebo | Pancrelipase
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Body Weight Composition
Description: Body weight composition will be determined at the time of accrual, and at 4 and 10 weeks of cross-over treatment.
Time Frame: Baseline, 4 weeks, 10 weeks
Population: Study was terminated due to difficulty in recruiting subjects. Data was not collected or analyzed.
Arm/Group | Placebo | Pancrelipase
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 10 weeks on all participants.
Arm/Group | Placebo | Pancrelipase
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT02985801/Prot_SAP_000.pdf